CLINICAL TRIAL: NCT03022708
Title: Prospective, Non-randomized, Pivotal Study to Assess the Safety and Efficacy of the Bioabsorbable Pulmonary Valved Conduit in Subjects Undergoing Right Ventricular Outflow Tract (RVOT) Reconstruction
Brief Title: Xeltis Bioabsorbable Pulmonary Valved Conduit Pivotal Study
Acronym: Xplore2
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xeltis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XEL-CR-03
Record Dates: First submitted 2017-01-10; First posted 2017-01-16 (Estimated); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Heart Defect, Congenital
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Xeltis Bioabsorbable Pulmonary Valved Conduit (Experimental): The Bioabsorbable Pulmonary Valved Conduit bio-absorbable, polymer-based medical device.
  The PV conduit is used in patients for correction or reconstruction of the Right Ventricular Outflow Tract (RVOT), in patients less than 22 years with any of the following congenital heart malformations:
  * Tetralogy of Fallot
  * Truncus Arteriosus
  * Pulmonary Atresia
  * Transposition of Great Arteries with Ventricular Septal Defect
  * Pulmonary Stenosis in combination with other defects in congenital heart defect (CHD) syndromes
  In addition, the PV conduit can be used for the following indications:
  * replacement of previously implanted, but dysfunctional, pulmonary homografts or valved conduits (except for mechanical valves, see exclusion criterion 3).
  * Patients undergoing a Ross procedure, where the PV conduit would replace the patient's own pulmonary valve which is used to replace a diseased aortic valve.
  Interventions: Device: Xeltis Bioabsorbable Pulmonary Valved Conduit

INTERVENTIONS:
Device: Xeltis Bioabsorbable Pulmonary Valved Conduit — Surgical implantation of Xeltis Bioabsorbable Pulmonary Valved Conduit

SUMMARY:
This is a multi-center prospective, single-arm, non-randomized, pivotal study that will continue to access the feasibility of the Xeltis Bioabsorbable Pulmonary Valved Conduit in subjects requiring right ventricular outflow tract correction or reconstruction due to congenital heart malformations.

ELIGIBILITY:
Inclusion Criteria:

1. Patient requiring RVOT reconstruction, suitable for 16 mm,18 mm, 20 mm and 22 mm valved conduit.
2. Male or Female.
3. Age > 2 years and < 22 years.
4. Right Ventricular to Pulmonary Artery peak gradient > 35mm Hg or moderate or severe Pulmonary regurgitation (≥3+), or have both (except for the patients undergoing a Ross procedure)
5. The patient, and the patient's parent / legal representative where appropriate, has been informed of the nature of the study, agrees to its provisions and has provided written informed consent by signing the approved informed consent form.
6. The patient, and the patient's parent / legal representative where appropriate, and the treating physician agree that the subject will return for all required post-procedure follow up visits and the subject will comply with clinical investigation plan required follow-up visits.

Exclusion Criteria:

1. Need for or presence of prosthetic heart valve at other position.
2. Need for concomitant surgical procedures (non-cardiac).
3. Patients with previously implanted pacemaker (including defibrillators), or mechanical valves.
4. Active infection or requiring current antibiotic therapy (if temporary illness, subject may be a candidate 4 weeks after discontinuation of antibiotics) or viral infection.
5. Active endocarditis.
6. Leukopenia, defined as White Blood cell Count < than:

   * 2-12 years: 5.0 ×103 /μL
   * 12 years - Adult:
   * Male: 4.5×103 /μL
   * Female: 4.5 ×103 /μL
7. Acute or chronic anemia, defined as Hemoglobin < than:

   * 2-12 years 11.5 g /dl
   * 12-18:
   * Male: 13 g /dl
   * Female 12 g /dl
   * Adult:
   * Male: 13.5 g /dl
   * Female: 12 g /dl Patients can be transfused to meet eligibility criteria
8. Thrombocytopenia, defined as Platelet count < than:

   * 150,000/mm3 Patients can be transfused to meet eligibility criteria
9. Severe chest wall deformity, which would preclude placement of the PV conduit.
10. Pulmonary hypertension (≥ half of systemic systolic pressure)
11. Right ventricular outflow tract aneurysm.
12. Known hypersensitivity to anticoagulants and antiplatelet drugs and to the device materials. .
13. Immunocompromised patient defined as: autoimmune disease, patients receiving immunosuppressant drugs or immune stimulant drugs.
14. Subject has chronic inflammatory / autoimmune disease.
15. Need for emergency cardiac or vascular surgery or intervention.
16. Major or progressive non-cardiac disease (liver failure, renal failure, cancer) that has a life expectancy of less than one year.
17. Currently participating, or participated within the last 30 days, in an investigational drug or device study.
18. Alcohol or drug abuse as defined by DSM IV-TR criteria for substance abuse - this includes the illicit use of cannabis within the last 12 months.
19. Pregnancy.
20. Females who are sexually active and are not willing to use adequate contraceptive precautions for the next 2 years
21. Subject has medical, social or psychosocial factors that, in the opinion of the Investigator, could impact safety or compliance.

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 56 (Estimated)
Dates: Start 2017-05-08 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Composite rate of events of device related death, re-operation or re-intervention at 12 months follow-up. | 12 months
  Measured once all 12 month follow up visits have been completed

SECONDARY OUTCOMES:
Overall rate of device related death due to device failure at 6 months follow up post implantation. | 6 months
  Measured once all 6 month follow up visits have been completed
Overall rate of mortality at 60 months follow up post implantation. | 60 months
  Measured once all 60 months follow up visits have been completed
Overall rate of subjects who require reoperation or re-intervention due to device failure 12 months. | 12 months
  Measured once all 12 month follow upvisits have been completed .
Overall rate of subjects with a mean pressure gradient across the area of conduit implantation of less than 40 mm Hg at 6 and 12 months follow up. | 6 and 12 months
  Measured by echography at 6 and 12 months follow up.
Overall rate of subjects with pulmonary regurgitation of equal or less than moderate at 6 and 12 months follow up. | 6 and 12 months
  Measured by echography at 6 and 12 months follow up.

OTHER OUTCOMES:
Measurement of growth of conduit in pediatric population measured at 6, 36, 48 and 60 months. A competent valve with increased valve diameter in age groups < 18 years in correlation with the increased body surface area. | Up to 60 months
  Measured with echocardiography at 6, 36, 48 and 60 months follow up.
Overall satisfaction of the implanting surgeon of the implantation procedure of the Bio-absorbable pulmonary valve conduit | Day 0 - Implant
  Measured with a questionnaire given to the implanting surgeon at the time of implantation of the pulmonary valve conduit.

CONTACTS AND LOCATIONS:
Overall Officials: Eliane Schutte, Study Director — Xeltis Inc
Locations (10):
- United States (7):
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Joe DiMaggio Children's Hospital, Hollywood, Florida
  - New York Presbyterian Hospital - Columbia University (Xplore1), New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Pittsburgh of UPMC (Xplore1), Pittsburgh, Pennsylvania
  - UTSW- Dallas Children's Hospital, Dallas, Texas
- Multiprofile Hospital for Active Treatment "National cardiology hospital" EAD, Department of Congenital Heart Defects Surgery, Sofia, Bulgaria
- Institut Jantung Negara Sdn Bhd, Kuala Lumpur, Malaysia
- University Children's Hospital of Cracow, Krakow, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Morales DL, Herrington C, Bacha EA, Morell VO, Prodan Z, Mroczek T, Sivalingam S, Cox M, Bennink G, Asch FM. A Novel Restorative Pulmonary Valve Conduit: Early Outcomes of Two Clinical Trials. Front Cardiovasc Med. 2021 Mar 4;7:583360. doi: 10.3389/fcvm.2020.583360. eCollection 2020. PMID 33748192